CLINICAL TRIAL: NCT05773209
Title: Effect of Repeated Low-level Red-light (RLRL) Therapy on the Choroid and the Retina in Diabetes and Diabetic Retinopathy
Brief Title: Choroidal and Retinal Changes After RLRL Therapy in Diabetes and Diabetic Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second People's Hospital of Foshan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SecondPeopleFoshan
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Retinopathy
Keywords: Repeated low-level red-light (RLRL) therapy; Choroidal thickness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RLRL of 100% intensity (Experimental): Participants will be treated with RLRL treatment (100% intensity) twice per day with an interval of at least 4 hours, each treatment last 3 minutes. Cross over arms after one month of use and one month of washout period.
  Interventions: Device: RLRL device
- RLRL of 5% intensity (Sham Comparator): Participants will be treated with the sham device (5% intensity) twice per day with an interval of at least 4 hours, each treatment last 3 minutes. Cross over arms after one month of use and one month of washout period.
  Interventions: Device: RLRL device

INTERVENTIONS:
Device: RLRL device — Crossover device (RLRL of 5% or 100% intensity - alternate to first group). Cross over arms after one month of use and one month of washout period.

SUMMARY:
The choroidal thickness was found to be thinner in diabetic eyes without retinopathy compared to healthy eyes, thus choroidal thickness might be an important parameter for the development of diabetic retinopathy in diabetic eyes without retinopathy. Repeated low-level red-light (RLRL) therapy is an emerging innovative and non-invasive treatment for a variety of eye diseases. Notably, RLRL was found to be effective in thickening choroidal thickness in a 1-year randomized controlled trial, indicating its potential in modulating blood flow in the fundus. This study aims to answer whether RLRL therapy can thicken choroidal thickness in adults with diabetes mellitus or diabetic retinopathy.

DETAILED DESCRIPTION:
The goal of this study is to investigate the effect of repeated low-level red-light (RLRL) therapy on the choroidal and retinal structures in diabetes mellitus and diabetic retinopathy. This study will be conducted with a prospective randomized cross-over design with a total follow-up of 3 months. The control group will use the sham device but with only 5% of the original device's power. Comprehensive ophthalmic examinations, including visual acuity, intraocular pressure, optical coherence tomography, optical coherence tomography angiography, slit lamp will be assesses at baseline and within the follow up

ELIGIBILITY:
Inclusion Criteria:

1. Aged 35-55 years
2. Diagnosis of type 2 diabetes mellitus
3. No DR or only mild non-proliferative DR (NPDR) assessed by baseline clinical ocular signs and 7-field fundus color photography

Exclusion Criteria:

1. Spherical equivalent (SE) ≤ -6.0 diopter or axial length ≥26 mm
2. Patients with complications such as DME and retinal detachment
3. History of ocular surgical operations
4. Severe systemic diseases
5. Those who could not cooperate with the examination for any reason
6. Cognitive impairment or mental illness
7. Patients with other ocular diseases

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in subfoveal choroidal thickness | 1 month
  Changes in subfoveal choroidal thickness after 1-month RLRL treatment, which is measured by optical coherence tomography.

SECONDARY OUTCOMES:
Changes in choroidal vascularity index | 1 month
  Changes in choroidal vascularity index after 1-month RLRL treatment, which is measured by optical coherence tomography.
Changes in OCTA-derived parameters of the choroid and retina | 1 month
  Changes in OCTA-derived parameters of the choroid and retina after 1-month RLRL treatment
Changes in DR grading | 1 month
  Changes in DR grading after 1-month RLRL treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Kong, PhD, Study Chair — The Second People's Hospital of Foshan, Guangdong Province,China

IPD SHARING:
Plan to Share IPD: No
Not Provided